CLINICAL TRIAL: NCT05996120
Title: Normothermic Versus Hypothermic Cardiopulmonary Bypass in Adult Cardiac Surgery: a Multicentre Feasibility Randomised Controlled Trial
Brief Title: Study on Optimal Temperature During Cardiopulmonary Bypass (THERMIC-4)
Acronym: THERMIC-4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: NHS National Waiting Times Centre Board (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Oxford University Hospitals NHS Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); University Hospitals Bristol and Weston NHS Foundation Trust (Other); University Hospitals, Leicester (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0910; IRAS (Other: 325522)
Record Dates: First submitted 2023-07-02; First posted 2023-08-16 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Heart Disease; Valvular Heart Disease; Cardiovascular Diseases; Surgery-Complications
Keywords: cardiopulmonary bypass; hypothermia; myocardial protection; neurologic protection
MeSH Terms: conditions — Myocardial Ischemia; Heart Valve Diseases; Cardiovascular Diseases; Hypothermia

STUDY DESIGN:
Intervention Model Description: Parallel group, open label, statistician blinded, multicentre, randomised controlled feasibility trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypothermic Cardiopulmonary Bypass (Active Comparator): Patients allocated to this arm will undergo standard care for coronary artery bypass grafting and/or valve surgery with mild hypothermia during CPB.
  Interventions: Procedure: Hypothermic Cardiopulmonary Bypass
- Normothermic Cardiopulmonary Bypass (Active Comparator): Patients allocated to this arm will undergo intervention care for coronary artery bypass grafting and/or valve surgery with normothermia hypothermia during CPB.
  Interventions: Procedure: Normothermic Cardiopulmonary Bypass

INTERVENTIONS:
Procedure: Hypothermic Cardiopulmonary Bypass — Mild hypothermia (between 32 - 35 °C) during cardiopulmonary bypass
  Arms: Hypothermic Cardiopulmonary Bypass
Procedure: Normothermic Cardiopulmonary Bypass — Normothermia (active maintenance of temperature between 36.5 °C to 37.5°C; no active cooling below 36.5 °C) during cardiopulmonary bypass
  Arms: Normothermic Cardiopulmonary Bypass

SUMMARY:
In order to perform heart surgery, a machine called cardiopulmonary bypass (CPB), or more commonly known as a heart-lung machine, is used to maintain the circulation of oxygenated blood needed by the rest of the body and its organs.

Historically, when a patient is connected to CPB, their body is cooled below the normal body temperature. This is known as hypothermia. This is because scientific studies have previously shown that reduced body temperature lowers metabolism and therefore offers more protection to the brain and other organs due to the reduced oxygen requirement. The evidence supporting this practice, however, has been challenged throughout the history of cardiac surgery, with studies supporting that normothermia, or normal body temperature, is a safe alternative. Despite this, the practice of hypothermia has persisted. Published data from a survey of 139 cardiac surgeons in the United Kingdom showed that 84% still routinely employ hypothermic CPB during surgery.

To assess whether normothermic or hypothermic CPB is safer, a clinical trial requiring a large sample size and high recruitment rates will be required. Therefore, the investigators aim to assess firstly the feasibility of trial recruitment and allocation adherence in this study. 100 adults across 10 different cardiac surgery centres in the United Kingdom will be recruited to a multicentre feasibility randomised controlled trial comparing normothermia (active comparator) against hypothermia (control comparator) during cardiopulmonary bypass in cardiac surgery. This study will also test the ability of the Cardiothoracic Interdisciplinary Research Network (CIRN), a trainee-led research collaborative, to collect pilot data on Major Adverse Cardiac and Cerebrovascular Events (MACCE) using a regulation-approved electronic application HealthBitⓇ. Participants will also be asked to complete quality of life surveys. The results of this study will subsequently inform a large, adequately powered randomised controlled trial for optimal temperature management during CPB.

DETAILED DESCRIPTION:
Primary Objective

To assess the feasibility of trial recruitment and delivery to target in the United Kingdom of a multicentre randomised controlled trial on normothermia versus hypothermia during cardiopulmonary bypass in adult cardiac surgery.

Secondary Objective

To assess the feasibility of conducting a multicentre randomized controlled trial (RCT) using a novel Good Clinical Practice (GCP) approved remote data capture as the primary trial database alongside analysis of routinely collected healthcare data.

To obtain pilot data, undertaken by the Cardiothoracic Interdisciplinary Research Network (CIRN), to inform a subsequent large, adequately powered RCT for optimal temperature management during CPB.

ELIGIBILITY:
INCLUSION CRITERIA

Participants may enter the trial if all of the following apply

1. Adult patients (≥ 18 years) scheduled for coronary artery bypass surgery and/or valve replacement/ repair, either in the elective or urgent setting.
2. European System for Cardiac Operative Risk Evaluation (EuroSCORE) II of 2 or higher.
3. Able to understand and communicate to provide informed consent.
4. Able to read and understand the English language.

EXCLUSION CRITERIA

Participants may not enter the trial if any of the following apply:

1. Patients undergoing coronary artery bypass surgery in combination with other procedures including cardiac or vascular procedures that require deep hypothermic arrest.
2. Patients undergoing emergency or salvage surgery.
3. Patients undergoing off-pump cardiac surgery.
4. Patients who are participating in another interventional trial.
5. Unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Total number of participants recruited over a 6 month period | 6 months
  The target recruitment rate is 1 participant per week per centre. The feasibility trial will be considered positive if 80% of target met, together with outcome 2.
Adherence rate to allocation | 6 months
  The feasibility trial will be considered positive if 74%* of target adherence to trial allocation is met, together with outcome 1.
  *74% is derived from 80% of target adherence of 92% as per Warm Heart Study

SECONDARY OUTCOMES:
Incidence of 6-week composite endpoint of Major Adverse Cardiac and Cerebrovascular Events (MACCE) | 6 weeks
  MACCE is defined as any post-operative death, stroke, new intra-aortic balloon pump insertion, new renal replacement therapy, re-operation and major bleeding in this feasibility trial.
Incidence of deep sternal wound infection, with or without treatment | 6 weeks
  Deep sternal wound infection is defined with at least one of the following criteria:
  (I) an organism is isolated from culture of mediastinal tissue or fluid (II) evidence of mediastinitis seen intraoperatively (III) presence of chest pain, sternal instability, or fever (> 38 °C), and purulent drainage from the mediastinum or isolation of organism present in a blood culture or from the mediastinal area.
Incidence of all adverse events | 6 weeks
  Composite of all reported adverse events. Examples of adverse events include: low cardiac output, suspected myocardial infarction, arrhythmias, infections, haemorrhage, and pulmonary embolus.
Critical care length of stay | 6 weeks
  Number of days a participant is admitted in cardiac critical care unit
Post-operative length of stay | 6 weeks
  Number of days a participant is an in-patient after index operation
Frequency of post-discharge healthcare resource utilisation | 6 weeks
  Number of visits to general practitioner (GP) and/or hospital, either district general hospital or tertiary hospital, will be recorded via HealthBitⓇ.
Quality of life post-operation: Medical Outcomes Study Short-Form 36 (SF-36) | 6 weeks
  Quality of life questionnaire (SF-36) will administered before surgery and at 6-week follow up
Quality of life post-operation: European Quality of Life-5 Dimensions (EQ-5D) | 6 weeks
  Quality of life questionnaire (EQ-5D) will administered before surgery and at 6-week follow up
Quality of life post-operation: World Health Organisation Disability Assessment Schedule (WHODAS) | 6 weeks
  Quality of life questionnaire (WHODAS) will administered before surgery and at 6-week follow up
Clinical Frailty Scale (CFS) post-operation | 6 weeks
  Clinical Frailty Scale will be recorded before surgery and at 6-week follow up

OTHER OUTCOMES:
Data completeness | 6 months
  Data recorded on HealthBitⓇ will be assessed for percentage of completion
Attrition rate | 6 months
  For ascertainment of the primary outcome and for planning of future large-scale study
User satisfaction of ResearchApp | 6 months
  Participants will be invited to complete optional survey on user satisfaction of ResearchApp

CONTACTS AND LOCATIONS:
Locations (11):
- United Kingdom (11):
  - Glenfield Hospital, University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Blackpool Victoria Hospital, Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Castle Hill Hospital, Hull University Teaching Hospitals NHS Trust, Cottingham
  - Golden Jubilee National Hospital, NHS Golden Jubilee, Glasgow
  - King's College Hospital, King's College Hospital NHS Foundation Trust, London
  - Royal Brompton Hospital, Guy's and St Thomas' NHS Foundation Trust, London
  - Harefield Hospital, Guy's and St Thomas' NHS Foundation Trust, London
  - John Radcliffe Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford
  - Derriford Hospital, Plymouth University Hospitals NHS Trust, Plymouth
  - Northern General Hospital, Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised individual participant data can be made available on request for future studies with ethics approval.
Supporting Information: Study Protocol, CSR
Time Frame: The investigators will retain the fully anonymised dataset indefinitely. The duration for which this will be shared will be determined on a case-by-case basis and defined in a Data Sharing Agreement.
Access Criteria: Requests must be from studies with appropriate ethics approval in place.